CLINICAL TRIAL: NCT02830451
Title: Metastatic Tumor Research and Outcome Network A Multicenter Prospective Registry for the Management and Outcome of Metastatic Spine Tumors
Brief Title: Metastatic Tumor Research and Outcomes Network
Acronym: MTRON
Status: Active, not recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Collaborators: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: MTRON
Record Dates: First submitted 2016-06-21; First posted 2016-07-12 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Spine Tumor
Keywords: Registry; Spine; Surgery; Medical Oncology; Radiation Oncology; Neoplasms; Metastasis; Chemotherapy; Radiation Therapy; Tumor Markers
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The registry aims to collect patient information such as patient demographics, co-morbidities, clinical, diagnostic, and therapeutic data, as well as information on adverse events and HRQOL outcomes specific for patients with metastatic spine tumor(s).

DETAILED DESCRIPTION:
To prospectively determine the prognostic variables (clinical, diagnostic, and therapeutic) within patients diagnosed with metastatic spine tumor(s) that are associated with:

* patient reported outcomes (HRQOL)
* morbidity data
* local tumor control
* survival

Outcome measures:

Variables which will be collected in the registry that are applicable to patients with metastatic spine tumor include:

* • Patient details
* Details of previous treatment
* Diagnosis
* Symptoms
* Treatment details for the index target
* Imaging information

The following outcome measures will be collected:

* Patient reported outcomes:

  * Euroqol EQ-5D-3L
  * Euroqol EQ-5D VAS - Quality of Life
  * Neck Pain Numeric Rating Scale (NRS)
  * Arm Pain NRS
  * Back Pain NRS
  * Leg Pain NRS
  * SOSGOQ
  * Patient assessment
* Ambulation
* Pain medication
* Nutritional Status Tool (PG-SGA©)
* Morbidity data
* Local disease recurrence data
* Overall survival data

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 or older.
* Patient diagnosed with a metastatic tumor of the spine
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the registry according to the Registry Plan
  * Signed and dated EC/IRB approved written informed consent (if consent is required by the EC/ IRB at the registry site)

Exclusion Criteria:

• Patient diagnosed with a primary tumor of the spine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with a metastatic tumor of the spine.
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient details | collected at baseline
  The following patient data will be collected:
  * gender, year of birth, height, weight, race
  * work status, education level, marital status
  * smoking, alcohol and recreational drug use
  * medication use
  * nutrition and vitamin intake
  * presence of osteoporosis
  * comorbidities according to the Charlson Comorbidity Index - CCI
Tumor details | collected at baseline, first prospective treatment and follow-up
  Primary cancer
  * Site of the primary cancer
  * Year of diagnosis
  * Status of the tumor (removed completely, partially, or not removed)
  * Signs of local control or tumor progression
  * Tumor subtype
  * Tumor markers
  Spine metastases
  * Date of initial diagnosis of spine metastases
  * Identification of index target
  * Vertebral location (i.e., C1, T3-T5, etc.)
  * Details of spine metastases and other metastases, if any
  * Activity of systemic metastases
  * Local control of metastatic tumor
  * Presence of pathologic fracture
  * Radiographic evidence of new spine metastatic disease
Symptoms | collected at baseline, first prospective treatment and follow-up
  For patients with metastatic spine tumor, it is important to understand the occurrence, location, and type of pain patients have at baseline and at follow-up visits. Pain symptoms assessed by the physician will therefore be collected in addition to the pain specific PROs.
  Bowel and bladder function will be assessed by the physician.
Treatment details - previous treatment of the index of the spine | Collected at baseline
  If the patient had previous treatment (surgery, radiation or systemic oncologic therapy) for the index target, the following information about the previous treatment will be collected at baseline:
  * Type(s) of treatment
  * Date(s) of treatment
  * Treated vertebrae level(s)
  * Procedure details
  * Hospital/center where the treatment was administered
  * ASIA impairment scale (applies only to previous surgical patients)
Imaging information | collected at baseline, first prospective treatment, discharge and at follow-up.
  Skeletal muscle and adipose tissue measurements will be made from CT scans. One transverse CT image of the inferior surface of L3 will be assessed by an independent assessor to calculate the visceral fat area to subcutaneous fat ratio (VFA/SFA ratio). This measurement will only be collected if the CT scan is according to standard of care and the method is described in a separate imaging manual. Additional CT scans will not be performed for this Registry.
  Imaging is critical to select the biopsy technique and for disease diagnosis. Follow-up imaging also plays an important role in monitoring disease status. Imaging data will be collected to serve as a data repository, so that images may be more easily retrieved later if necessary.
  Imaging data
  * Image type (e.g. MRI, CT, PET, etc.)
  * Date taken
  * Name of institution storing image
Patient reported outcomes - Euroqol EQ-5D-3L / - EQ-5D VAS | collected at baseline, first prospective treatment, discharge and at follow-up.
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Ambulation | collected at baseline, discharge and at follow-up.
  Details about the ability of the patient to walk, cause of ambulation loss, use of an assistive device, and timing will be collected.
  10 meter walk test (10 MWT) If the patient is able to ambulate without physical assistance (i.e. without help of a person), ambulation will be assessed by the 10MWT (walking aids are allowed). The 10MWT evaluates the time required to walk 10 meters. Patients should walk 10 meters with 2 meters for acceleration and deceleration. The patient will be timed from when the patient's toes of the leading foot cross the 2 meter line to when the patient's toes of the leading foot cross the 8 meter line. The test should be performed three times and the results will be averaged. The patient should be instructed to perform the test at a comfortable walking pace.
Nutritional status tool | collected at baseline, first prospective treatment, discharge and at follow-up.
  The Scored Patient-Generated Subjective Global Assessment (PG-SGA©) sets the standard of and is the preeminent interdisciplinary patient assessment (weight, intake, symptoms, functional status, disease state, metabolic stress and nutritional physical examination) in oncology and other chronic catabolic conditions.
  The Scored PG-SGA© includes the four patient-generated historical components ('Weight History', 'Food Intake', 'Symptoms' and 'Activities and Function'), the professional part (Diagnosis, Age, Metabolic stress, and Physical Exam), the Global Assessment (A = well nourished, B = moderately malnourished or suspected malnutrition, C = severely malnourished), the total numerical score, and nutritional triage recommendations. Subsequently, the Scored PG-SGA© allows for triaging of specific nutrition interventions, as well as facilitating quantitative outcomes data collection.
  This assessment is available in a variety of languages and as a metric as well as a non-metric version.
Morbidity data - Adverse events | collected at first prospective treatment, discharge and at follow-up.
  * related to surgery Intra- and postoperative complication data will be recorded for all surgically treated patients during the standard of care scheduled follow-up visits. Complications will be assessed by evaluating the patient's medical files from the time treatment was initiated until the day of follow-up. The Spine AdVerse Events Severity system, version 2 (SAVES V2) AE abstraction tool will be used to record the morbidity data.
  * related to radiation and/or systemic oncologic therapy
  For patients treated with RT and/or systemic oncologic therapy, complications and severity grade related to the treatment will be recorded during the standard of care scheduled follow-up visits according to a predefined list:
  The predefined list and severity grading system are according to the National Cancer Institute Guidelines.
Local disease recurrence data | collected at baseline and at follow-up.
  At every FU visit, each patient, regardless of which stage they are at in their treatment, will be evaluated for local disease control. Presence or absence of local control and distant metastases should be confirmed through imaging. The timing of the assessment will be performed in accordance with local standard of care scheduled FU visits.
Survival | collected at first prospective treatment, discharge and at follow-up.
  FU visits will be scheduled and performed according to the local standard of care and at each scheduled visit the patient's survival will be documented. In case a patient misses a scheduled visit it will be assessed if the patient is still alive.
Treatment details - Current treatment of the index target of the spine | collected at first prospective treatment and at follow-up.
  Since there is a spectrum of different treatment options and combinations for patients with a metastatic spine tumor, detailed information about the three main treatment options (surgery, radiation, and systemic oncologic therapy) for the index target will be collected. The treatment intent, including administration (primary, neo-adjuvant, and adjuvant) will also be collected.
Treatment details - Current treatment for the primary cancer | collected at baseline, first prospective treatment and at follow-up.
  Information on the status of the primary cancer as well as on ongoing treatment of the primary cancer will be collected at baseline and at follow-up.
Patient reported outcomes - Pain Numeric Rating Scale | collected at baseline, first prospective treatment, discharge and at follow-up.
  The Pain NRS is an 11-point scale where the end points are the extremes of no pain (0 points), or worst imaginable pain (10 points). It measures subjective intensity of pain and the patient rates his/her overall or average daily pain.
Patient reported outcomes - Spine Oncology Study Group Outcome Questionnaire (SOSGOQ) | collected at baseline, first prospective treatment, discharge and at follow-up.
  This is a new HRQOL outcome tool which was developed specifically for metastatic spine tumor. It is currently available in English and Hungarian. It contains 20 items representing all four domains of the International Classification of Function and Disability. Additionally there are seven follow-up questions referring to treatment satisfaction. It is made up of five domains: physical function, neural function, pain, mental health and social function. It was developed as a comparison to the SF-36 for patients with spine tumors.

SECONDARY OUTCOMES:
Symptoms: American Spinal Injury Association (ASIA) Impairment Scale | collected at baseline, first prospective treatment, discharge and at follow-up.
  International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) ISNCSCI is a standardized examination to determine neurologic function and has been a standard clinical assessment for patients with neurological deficit. The modified ISNCSCI used in this study will assess the Motor Score and the American Spinal Injury Association (ASIA) Impairment Scale
Symptoms: Eastern Cooperative Oncology Group (ECOG) classification | collected at baseline, first prospective treatment, and at follow-up.
  The ECOG developed a scale from 0 to 5 to assess the patient's disease progression and how the disease affects the patient's daily living abilities (9). The lower the score the better the status of the patient, being 0 fully active and 5 dead.
Symptoms: Epidural Compression Classification | Collected at baseline
  The Spine Oncology Study Group developed and validated a 6-point grading system to describe the degree of epidural spinal cord compression based on axial T2-weighted MR images at the site of most severe compression. This assessment can be used to help guide treatment and can serve as a classification scheme.
Spine Instability Neoplastic Score (SINS) | collected at baseline and first prospective treatment,
  The SOSG developed and validated a classification system to assist clinicians in defining tumor-related instability. It is assessed by adding together six individual component scores: spine location, pain, lesion bone quality, radiographic alignment, vertebral body collapse, and posterolateral involvement of the spinal elements. SINS has demonstrated clinically acceptable reliability among surgeons, radiation oncologists, and radiologists. The total SINS score can range from a score of 0 to 18. The total score has been divided into three categories of stability: stability (score of 0-6), indeterminate instability (score of 7-12), and instability (score of 13-18). Surgical consultation is recommended for patients with SINS scores ≥ 7. SINS will be assessed at baseline and/or prior to first prospective treatment. The most severe lesion within the index target should be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Charles G. Fisher, MD, Principal Investigator — Vancouver General Hospital and the University of British Columbia
Locations (25):
- United States (11):
  - University of California The UCSF Spine Center Department of Neurological Surgery, San Francisco, California
  - Rush University Medical Center University Neurosurgery, Chicago, Illinois
  - Johns Hopkins University Department of Neurosurgery / Spine Division, Baltimore, Maryland
  - Harvard Medical School Department of Neurosurgery, Boston, Massachusetts
  - Mayo Clinic Department of Neurosurgery, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester School of Medicine and Dentistry Department of Orthopaedic Surgery and Neurosurgery, Rochester, New York
  - Westchester Medical Center Department of Neurosurgery, Valhalla, New York
  - Penn Presbyterian Medical Center Department of Neurosurgery, Philadelphia, Pennsylvania
  - The Warren Alpert Medical School of Brown university Department of Neurosurgery, Providence, Rhode Island
  - The University of Texas MD Anderson Cancer Center Department of Neurosurgery, Houston, Texas
- Monash University Melbourne, Clayton, Victoria, Australia
- Canada (5):
  - Vancouver General Hospital and the University of British Columbia, Vancouver, British Columbia
  - Winnipeg Spine Program University of Manitoba Department of Surgery, Winnipeg, Manitoba
  - Toronto Western Hospital Department of Neurosurgery Division of Surgery, Toronto, Ontario
  - University of Toronto Odette Cancer Centre - T2 158 Sunnybrook Health Sciences Ccenter, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Universitätsklinikum Carl Gustav Carus der Technischen Universität Dresden, Dresden, Saxony, Germany
- National Center for Spinal Disorders and Buda Health Center, Budapest, Hungary
- Italy (2):
  - Instituto Ortopedico Rizzoli Department of Oncologic and Degenerative Spine Surgery, Bologna, Emilia-Romagna
  - IRCCS Istituto Ortopedico Galeazzi Centro die Chirurgia Ortopedica Oncologica e Ricostr, Milan, Lombardy
- Kanazawa Medical University Hospital Department of Orthopaedic Surgery, Uchinoda, Ishikawa-ken, Japan
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- National University of Singapore Department of Orthopaedic Surgery, Singapore, Singapore
- Universitätsspital Basel Wirbelsäulenzentrum, Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No